CLINICAL TRIAL: NCT02982434
Title: Injection of the New Pharmaceutical Composition Containing Botulinum Toxin Into Epicardial Fat Pads to Treat Atrial Fibrillation After Coronary Artery Bypass Grafting
Brief Title: The New Pharmaceutical Composition Containing Botulinum Toxin to Treat Atrial Fibrillation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RSTD_021216
Record Dates: First submitted 2016-12-01; First posted 2016-12-05 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-12

CONDITIONS: Atrial Fibrillation; Ischemic Heart Disease
Keywords: atrial fibrillation; botulinum toxin; ischemic heart disease
MeSH Terms: conditions — Atrial Fibrillation; Myocardial Ischemia | interventions — Saline Solution; Coronary Artery Bypass

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Group 1 (Experimental): All patients underwent conventional CABG surgery. After the main stage of the surgery new pharmaceutical composition containing botulinum toxin (50 U/1 mL) was injected into the entire four visible area of the major epicardial fat pads. First epicardial left atrial fat pad is located anterior to the right superior pulmonary vein and corresponding to the anterior right ganglionated plexi (GP); second epicardial fat pad is located inferoposterior to the right inferior pulmonary vein and corresponding to the inferior right GP; third fat pad is located anterior to the left superior pulmonary vein (PV) and left inferior PV (between the PVs and left atrial appendage (LAA), corresponding to the Marshall tract GP and superior left GP; forth fat pad located inferiorly to the left inferior PV and extends posteriorly and corresponding to the inferior left GP
  Interventions: Drug: Pharmaceutical composition containing botulinum toxin; Procedure: Coronary artery bypass grafting
- Group 2 (Active Comparator): All patients underwent conventional cardiac surgery. After the main stage of the surgery 0.9% normal saline (1 mL at each fat pad) was injected into the entire four visible area of the major epicardial fat pads. First epicardial left atrial fat pad is located anterior to the right superior pulmonary vein and corresponding to the anterior right GP; second epicardial fat pad is located inferoposterior to the right inferior pulmonary vein and corresponding to the inferior right GP; third fat pad is located anterior to the left superior PV and left inferior PV (between the PVs and LAA), corresponding to the Marshall tract GP and superior left GP; forth fat pad located inferiorly to the left inferior PV and extends posteriorly and corresponding to the inferior left GP
  Interventions: Drug: 0.9% normal saline; Procedure: Coronary artery bypass grafting

INTERVENTIONS:
Drug: Pharmaceutical composition containing botulinum toxin
  Arms: Group 1
Drug: 0.9% normal saline
  Arms: Group 2
Procedure: Coronary artery bypass grafting

SUMMARY:
The aim of this prospective randomized double-blind study was to compare the efficacy of new pharmaceutical composition containing botulinum toxin injection in epicardial fat pads for preventing recurrences of atrial tachyarrhythmia in patients with paroxysmal atrial fibrillation undergoing coronary artery bypass grafting.

ELIGIBILITY:
Inclusion Criteria:

* Patients with paroxysmal AF (recurrent episodes for at least 2 years, with ≥ 6 episodes over the last 6 months)
* At least one failed antiarrhythmic drug
* Indication for cardiac surgery (e.g. coronary artery bypass grafting, valve repair/replacement) according to the American College of Cardiology/American Heart Association (ACC/AHA) guidelines for cardiac surgery

Exclusion Criteria:

Previous heart surgery or atrial fibrillation ablation procedure Emergency coronary artery bypass grafting Unstable angina or heart failure Persistent atrial fibrillation or atrial fibrillation at the time of screening Planned maze procedure or pulmonary vein isolation Unwillingness to participate

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-12 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Freedom from any atrial tachyarrhythmias | 12 months
  Recurrence of >30 s of any atrial tachyarrhythmia, including atrial fibrillation and atrial flutter/tachycardia, after cardiac surgery procedure with no antiarrhythmic drug

SECONDARY OUTCOMES:
number of deaths | 12 month
time intervals from end of surgery to weaning from ventilation, extubation and discharge from ICU | 1 month
incidence of congestive heart failure | 12 month
incidence of sustained ventricular arrhythmias | 12 month
stroke or transient ischemic attack | 12 month
incidence of myocardial infarction | 12 month
rehospitalization | 12 months

CONTACTS AND LOCATIONS:
Locations (2):
- Russia (2):
  - State Research Institute of Circulation Pathology, Novosibirsk
  - Cardiology Research Institute, Tomsk